CLINICAL TRIAL: NCT00363480
Title: Asthma Control Assessment Via ACT and DRC in Asthmatics Treated With Seretide (50/250) Over 12 Weeks
Brief Title: Results Of Patient Rated Asthma Control Test In Comparison To Diary Card Data
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAM 106538
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: Asthma; Asthma Control Test; SERETIDE
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Fluticasone; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SFC 50/250 mcg (Experimental): Participants received the combination product, fluticasone 250 microgram (mcg) plus salmeterol 50 mcg (SFC 50/250 mcg) for 12 weeks. Study treatment was received using DISKUS™ powder inhalers, one dose in morning and evening. Study medication was dispensed at visits 3, 4, and 5 for 30 days each. The participants were provided with salbutamol rescue medication if they developed acute asthmatic symptoms. This medication was provided in metered dose inhalers containing at least 200 puffs of 100 mcg salbutamol. Use of rescue medications was recorded in the participant's asthma diaries. Stable dosages of other concomitant medications were allowed if they had no impact on the outcome criteria.
  Interventions: Drug: Salmeterol/Fluticasone 50/250 mcg; Drug: Salbutamol 100 mcg; Device: DISKUS™ powder inhalers

INTERVENTIONS:
Drug: Salmeterol/Fluticasone 50/250 mcg — Participant received salmeterol/fluticasone combination 50/250 mcg using DISKUS™ powder inhalers.
Drug: Salbutamol 100 mcg — This medication was provided in metered dose inhalers containing at least 200 puffs of 100 mcg salbutamol.
Device: DISKUS™ powder inhalers — Participant received salmeterol and fluticasone using DISKUS™ powder inhalers.

SUMMARY:
The majority of asthma patients are not well controlled, despite the availability of asthma medication that could effectively treat the disease. In this study uncontrolled patients who are steroid-naive or on low dose inhaled corticosteroids will be treated with Seretide (salmeterol/fluticasone combination, SFC) 50/250 µg twice daily. The asthma control test (ACT) will be used to detect differences in the level of asthma control during treatment. The study aims to show a correlation between improvements of ACT und the level of asthma control which will be reached by the patients.

The aim of the study is to show that most of symptomatic asthma patients can reach 'well controlled asthma' with SFC. We get information about ACT in daily practice and physicians are trained to use the asthma control test as a screening tool and for follow up of asthma management. Correlations are expected between the improvements in ACT, Quality of Life and asthma control according to the Gaining Optimal Asthma controL (GOAL) criteria.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of asthma
* Reversibility >12% after inhalation of 200 µg Salbutamol
* willingness and ability to complete daily record card on daily basis and to measure morning PEF on daily basis
* 80% compliance in diary card completion asthma control status: Uncontrolled based on the GOAL criteria

Exclusion criteria:

* Change of asthma medication during the last 4 weeks
* Asthma exacerbation characterized by use of oral corticoids during the last 3 months Pretreatment with inhaled corticosteroids more than 500 mcg Beclometasondipropionat or equivalent per day or other controller therapy during the last 3 months
* upper or lower respiratory tract infection during the RUN-IN period moderate or severe asthma exacerbation during the RUN-IN period
* Non compliance with use of Discus, PEF-meter and incomplete diary card data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2006-05-17 (Actual); Primary Completion 2007-09-01 (Actual); Study Completion 2007-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- Germany (23):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Kaufbeuren, Bavaria
  - GSK Investigational Site, Landsberg am Lech, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Uttenreuth, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Wedel, Hamburg
  - GSK Investigational Site, Bad Arolsen, Hesse
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Braunschweig, Lower Saxony
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Greiz, Thuringia
  - GSK Investigational Site, Sonneberg, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 27 centers in Germany from 17 May 2006 to 6 September 2007 on participants diagnosed with perennial bronchial asthma.
Pre-assignment Details: A total of 261 participants were screened, of which 40 were screen failure, remaining 221 participants entered the treatment period.
Period: Overall Study
Arm/Group | SFC 50/250 mcg
Started | 221
Completed | 204
Not Completed | 17
Not completed — Criteria for treatment period not fulfil | 1
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 5
Not completed — Non-compliance of subject | 1
Not completed — Participant discontinued on its own | 1

BASELINE CHARACTERISTICS:
Groups:
- SFC 50/250 mcg: Participants received SFC 50/250 mcg for 12 weeks. Study treatment was received using DISKUS powder inhalers, one dose in morning and evening. Study medication was dispensed at visits 3, 4, and 5 for 30 days each. The participants were provided with salbutamol rescue medication if they developed acute asthmatic symptoms. This medication was provided in metered dose inhalers containing at least 200 puffs of 100 mcg salbutamol. Use of rescue medications was recorded in the participant's asthma diaries. Stable dosages of other concomitant medications were allowed if they had no impact on the outcome criteria.
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Well Controlled Participants as Per Gaining Optimal Asthma Control (GOAL) Criteria After 12 Week Compared to Percentage of Participants With Asthma Control Test (ACT) Score of 20-25 for Week 9 to Week 12
Description: A week with well controlled asthma, when two or more of the criteria were fulfilled (diary entries): At most 2 days per week with 24-hour symptom score >1 (Range: 0= None to 5= severe), rescue salbutamol use on <= 2 days and at most 4 occasions per week, and a morning peak flow >= 80% of the predicted value on each day per week. All of the criteria which includes no night-time awakenings due to asthma (diary entry), no emergency visits (diary entry), no exacerbations and no treatment-related adverse events leading to treatment change are fulfilled. The total ACT score is based on a range of 5 to 25. Higher score indicates better asthma control. A score of 19 or less may be a sign that asthma symptoms are not under control.
Time Frame: Week 9 to Week 12
Population: Modified Intent-to-Treat population, participants covering treatment period of at least 8 weeks and with assessable asthma control at the end of the treatment period by both criteria (GOAL, ACT), and without major protocol deviations. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Percentage
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 170
Percentage
  GOAL | 33.5
  ACT | 64.1
Statistical Analysis 1: Comparison: SFC 50/250 mcg; Comparison between GOAL and ACT response; Test type: Superiority or Other; p < 0.0001, McNemar; Percentage diffrence = -30.6, 95% CI 2-sided [-37.89 to -23.29]

2. Secondary Outcome: Change From Baseline in Percentage of Participants With ACT Score of 20-25 at Week 12
Description: The total ACT score is based on a range of 5 to 25. Higher score indicates better asthma control. A score of 19 or less may be a sign that asthma symptoms are not under control. In order to derive the total ACT score, all 5 questions needed to be answered. Change from baseline value was calculated by subtracting baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Baseline (Visit 3) and Week 12
Population: Full Analysis Set comprised of all participants with at least one post-baseline (Visit 3) efficacy measurement during clinic visits (Visit 4, 5, 6) or valid diary data documented for at least one week post-baseline was included. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 213
Participants
  Baseline | 32
  Week 12 | 139
Statistical Analysis 1: Comparison: SFC 50/250 mcg; Test type: Superiority or Other; t-Distribution = 50.2, 95% CI 2-sided [43.15 to 57.32]

3. Secondary Outcome: Change From Baseline in Mean ACT Score at Visit 6
Description: The total ACT score is based on a range of 5 to 25. Higher score indicates better asthma control. A score of 19 or less may be a sign that asthma symptoms not under control. In order to derive the total ACT score, all 5 questions had to be answered. Change from baseline value was calculated by subtracting baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Baseline (Viait 3) and Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 203
Score on a scale | 5.0 (4.3)

4. Secondary Outcome: Number of Participants With Well Controlled and Totally Controlled Asthma at Week 12
Description: Well controlled or totally controlled asthma assessments were done according to the GOAL criteria. A week with well controlled asthma, when two or more of the criteria were fulfilled (diary entries): At most 2 days per week with 24-hour symptom score >1(Range: 0= None to 5= severe), rescue salbutamol use on <= 2 days and at most 4 occasions per week, and morning peak flow >= 80% of the predicted value on each day per week. All of the criteria which included no night-time awakenings due to asthma (diary entry),no emergency visits (diary entry), no exacerbations and no treatment-related adverse events leading to treatment change were fulfilled. The total ACT score was based on a range of 5 to 25. Higher score indicates better asthma control. A score of 19 or less may be a sign that asthma symptoms are not under control. Change from baseline value was calculated by subtracting baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 217
Participants
  Well Controlled | 65 [23 to 36]
  Totally Controlled | 29

5. Secondary Outcome: Change From Baseline in Quality of Life Using the Asthma Quality of Life Questionnaire (AQLQ)
Description: For the level of asthma control, baseline values were derived taking the last 8 weeks during the pre-treatment period prior to Visit 3 into consideration. Regarding derived variables based on the asthma diary, data from the last week prior to Visit 3 was taken. Visit 3, regarded as baseline. AQLQ has 32 questions regarding activities, emotions, symptoms, and environmental triggers. Each item values range from 1 (maximum impairment) to 7 (no impairment). A positive change from baseline score indicates improvement.
Time Frame: Baseline (Visit 3) up to Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 188
Score on Scale | 0.83 (0.91)

6. Secondary Outcome: Correlation of Change in AQLQ Score and Change in ACT Score
Description: Correlation between change in the AQLQ and ACT score was tabulated using the Pearson coefficient of correlation (linear correlation). The AQLQ contained 32 items in 4 domains: activity limitation, symptoms, emotional function and environmental stimuli. Scores for the domains as well as the overall score were scaled within a range of 1 (worst) to 7 (best).
Time Frame: Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 217
participants | 0.522

7. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) to Week 12
Description: FEV1, an amount of air exhaled by a person during a forced breath in one second. FEV1 assessed at Visit 1 and at Visits 3, 4, 5, 6. Baseline was the measurement at Visit 3. Change from baseline value was calculated by subtracting baseline value from week 12 value.
Time Frame: Baseline (Visit 3) up to Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Litre/second (L/Sec)
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 217
Litre/second (L/Sec)
  Week 4 | 0.133 (0.320)
  Week 8 | 0.212 (0.359)
  Week 12 | 0.181 (0.372)

8. Secondary Outcome: Change From Baseline in Mean Morning Percent Predicted Peak Expiratory Flow (PEF) at Week 12
Description: PEF, a person's maximum speed of expiration, as measured with a peak flow meter, a small, hand-held device used to monitor a person's ability to breathe out air. The mean morning PEF evaluated by means of the data documented in the asthma diaries. Change from baseline value was calculated by subtracting baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Baseline (Visit 3) and Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 194
Percentage | 7.798 (10.302)

9. Secondary Outcome: Change From Baseline in Mean 24-hour Symptom Score at Week 12
Description: The various symptoms like wheezing, shortness of breath, coughing and chest tightness were assessed by the participants every morning using a symptom score scale which ranged from 0 (no symptoms during the past 24 hours) to 5 (symptoms so severe that participant could not go to work or carry out other normal daily activities). Change from baseline value was calculated by subtracting baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Baseline (Visit 3) and Week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 191
Score on Scale | -0.590 (0.948)

10. Secondary Outcome: Change From Baseline in Number of Additional Usage of Salbutamol at Week 12
Description: Salbutamol was given as a rescue medicine, used on <= 2 days and at most 4 occasions per week. Change from baseline value was calculated by subtracting the baseline value from week 12 value. The assessments recorded at Visit 3 were considered as Baseline assessments.
Time Frame: Baseline (Visit 3) and week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of occassions
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 190
Number of occassions | -0.933 (1.331)

11. Secondary Outcome: Percent Change From Baseline in Number of Nights With no Nocturnal Awakening at Week 12
Description: Number of nights with no night time awakening were recorded at Week 12. Baseline was the last corresponding time period immediately prior to Visit 3.
Time Frame: Baseline (Visit 3) and week 12
Population: Full Analysis Set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 182
Percent Change | 7.228 (24.921)

12. Secondary Outcome: Number of Participants With Emergency Visits Due to Asthma
Description: Frequencies of emergency visits per participant were recorded during treatment period. Only the participants at risk were considered when calculating the incidence rates.
Time Frame: Up to week 12
Population: Safety set comprised of participants who received study medication at least once s participants who did not administer any study medication (those who returned all study medication dispensed) were not included in the Safety Set. Only those participants available at the indicated time points were analyzed.
Measure: Number; unit: Participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 202
Participants
  At least 1 day | 13
  1 day | 10
  2 days | 2
  3-4 days | 1
  5-9 days | 0

13. Secondary Outcome: Number of Participants With Adverse Events (AE) Leading to a Change in Asthma Treatment
Description: AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. Number of participants with AE who lead to change in asthma treatment were reported.
Time Frame: Up to Week 12
Population: Safety Set.
Measure: Number; unit: Participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
Participants | 4

14. Secondary Outcome: Assessment of Tolerability by Number of Participants With at Least One Treatment Emergent Serious and, Non-serious AE
Description: An AE is any untoward medical occurrence in a participant or clinical AE was any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which did not necessarily have a causal relationship with the treatment. Number of participants with at least one treatment emergent serious and, non-serious AE were reported.
Time Frame: Up to Week 12
Population: Safety Set.
Measure: Number; unit: Participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
Participants
  Any Non-Serious AE | 76
  Any Serious AE | 1

15. Secondary Outcome: Assessment of Tolerability by Change From Baseline of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were recorded over time (Visit 1, 3, 4, 5, and 6). Baseline was the measurement at Visit 3. Change from baseline value was calculated by subtracting baseline value from week 12 value.
Time Frame: Baseline (Visit 3) up to Week 12
Population: Safety Set. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
millimeters of mercury (mmHg)
  SBP, Week 4: number analyzed (Participants) | 212
  SBP, Week 4 | 0.8 (12.7)
  SBP, Week 8: number analyzed (Participants) | 205
  SBP, Week 8 | -0.7 (11.3)
  SBP, Week 12: number analyzed (Participants) | 203
  SBP, Week 12 | 0.2 (13.5)
  DBP, Week 4: number analyzed (Participants) | 212
  DBP, Week 4 | 0.2 (8.8)
  DBP, Week 8: number analyzed (Participants) | 205
  DBP, Week 8 | -0.2 (8.4)
  DBP, Week 12: number analyzed (Participants) | 203
  DBP, Week 12 | 0.6 (9.0)

16. Secondary Outcome: Assessment of Tolerability by Change From Baseline of Pulse Rate
Description: Pulse rate was recorded over time (Visit 1, 3, 4, 5, and 6). Baseline was the measurement at Visit 3. Change from baseline value was calculated by subtracting baseline value from week 12 value.
Time Frame: Baseline (Visit 3) up to Week 12
Population: Safety Set. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
Beats per minute (bpm)
  Week 4: number analyzed (Participants) | 212
  Week 4 | 1.0 (9.0)
  Week 8: number analyzed (Participants) | 205
  Week 8 | -0.2 (9.1)
  Week 12: number analyzed (Participants) | 203
  Week 12 | 0.6 (10.2)

17. Secondary Outcome: Number of Participants With Occurrence of (Near-) Incidents Associated With Peak Flow Measurements
Description: Frequencies of participants with at least one (near-) incident associated with peak flow measurements were recorded. analysis was done on safety population.
Time Frame: Up to Week 12
Population: Safety Set.
Measure: Number; unit: participants
Arm/Group | SFC 50/250 mcg
Number analyzed (Participants) | 221
participants | 0

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: The AE and SAEs were recorded using safety set of population.
Arm/Group | SFC 50/250 mcg
All-Cause Mortality (participants affected / at risk) | 1/221
Serious Adverse Events (participants affected / at risk) | 1/221
Other Adverse Events (participants affected / at risk) | 76/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SFC 50/250 mcg (N=221)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SFC 50/250 mcg (N=221)
Angina pectoris (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Gingivitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Local swelling (General disorders) | 1
Chest pain (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Gastrointestinal infection (Infections and infestations) | 1
Borrelia infection (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 6
Bronchitis (Infections and infestations) | 12
Nasopharyngitis (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Epicondylitis (Injury, poisoning and procedural complications) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Blood uric acid increased (Investigations) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 23
Sleep disorder (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.